CLINICAL TRIAL: NCT00994526
Title: Effect of Processed Meat on Colorectal Carcinogenesis. Study of Mechanisms. Choice of Preventive Strategies
Brief Title: Processed Meat and Colon Carcinogenesis
Acronym: Hemcancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Principal Investigator, Nathalie Meunier, Clinical research Assistant, University Hospital, Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AU794; IDRCB 2009-A00322-55 (Registry Identifier: Afssaps); 04/2009 FPIERRE (Other: CRNH)
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Processed meat; Calcium; Vitamin E; Preventive strategies
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ATF7IP protein, human; Calcium; Vitamin E

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ham (Placebo Comparator)
  Interventions: Other: Ham
- Ham + calcium (Experimental)
  Interventions: Other: Ham + calcium
- Ham + vitamin E (Experimental)
  Interventions: Other: Ham + vitamin E

INTERVENTIONS:
Other: Ham — Ham : 180 g per day during 4 days
  Arms: Ham
Other: Ham + calcium — Ham : 160g/d during 4 days calcium : 1000mg/d during 4 days
  Arms: Ham + calcium
Other: Ham + vitamin E — Ham : 160g/d during 4 days Vitamin E : 80 mg/d during 4 days
  Arms: Ham + vitamin E

SUMMARY:
Colorectal cancer kills forty five people in France every day. Epidemiological studies suggest that two cases out of three could be prevented and show that processed meat intake is a consistent risk factor. The aim of this study is to understand how meat promotes cancer, to find protective strategies, and to make compelling dietary recommendations.

DETAILED DESCRIPTION:
18 healthy volunteers will be randomized and will start the study. The study will last 4 weeks for each subject. The first week will be a week of adaptation (or run-in period) to the diet which they will have to follow for the duration of study. During this period, they will collect 2 samples of stools and urine. Then subjects will alternate 4 days of diet either with ham, or with ham and calcium, or with ham enriched with vitamin E. At least, 3 days will separate every period (wash-out) of nutritional intervention. Urines and stools will be collected last 3 days of every interventional period and also last day of every wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Body mass index 20 <= BMI <= 30 kg/m2
* Affiliated to French National Health Insurance
* Subject giving his written informed consent
* Subject considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* Positive serologies to HIV or HCV, determined on blood samples
* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Previous familial of colon, ovarian or breast cancer
* Chronic pathologies : cardiovascular diseases, cancer, chronic inflammation diseases, renal, intestinal impairments
* Dislike ham
* Heavy consumer of alcohol
* Practising intensive physical exercise
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Dietary habits unreliable to controlled food intake
* Being in exclusion on the National Volunteers Data file

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Urinary biomarker (DHN-MA:dihydroxynonene mercapturic acid), will be measured before and after every interventional period | Twice a week, before and after every 4 days of interventional period

SECONDARY OUTCOMES:
Fecal biomarkers | twice a week, before and after every 4 days of interventional period

CONTACTS AND LOCATIONS:
Overall Officials: Noël Cano, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand; Fabrice Pierre, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre de Recherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pierre FH, Martin OC, Santarelli RL, Tache S, Naud N, Gueraud F, Audebert M, Dupuy J, Meunier N, Attaix D, Vendeuvre JL, Mirvish SS, Kuhnle GC, Cano N, Corpet DE. Calcium and alpha-tocopherol suppress cured-meat promotion of chemically induced colon carcinogenesis in rats and reduce associated biomarkers in human volunteers. Am J Clin Nutr. 2013 Nov;98(5):1255-62. doi: 10.3945/ajcn.113.061069. Epub 2013 Sep 11. PMID 24025632
- See also: Related Info — http://www.inra.fr